CLINICAL TRIAL: NCT04318665
Title: Early Diagnosis of Mortality Using Admission CT Perfusion in Severe Traumatic Brain Injury Patients (ACT-TBI Study)
Acronym: ACT-TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jai Shankar, Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS23683 (B2020:018)
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Traumatic Brain Injury
Keywords: TBI, CTP
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT Perfusion (Experimental): Severe TBI patients will be undergoing CT perfusion test
  Interventions: Diagnostic Test: CT Perfusion

INTERVENTIONS:
Diagnostic Test: CT Perfusion — Severe Traumatic Brain Injury patients will be undergoing CT perfusion test

SUMMARY:
Background: Severe traumatic brain injury (TBI) is a principal cause of post-injury hospitalization, disability, and death throughout the world. TBI is the leading cause of death and disability among young healthy people under 45 years of age and is predicted to be the most prevalent and costliest neurological condition in Canada through the year 2031.

TBI is commonly classified into mild, moderate, and severe categories using the Glasgow Coma Scale (GCS), with "severe TBI" defined as a GCS score ≤ 8. Severe TBI is a clinical emergency, during which the trauma team works swiftly to provide the appropriate care. Outcome assessment after TBI is complex and is influenced by pre-injury and injury factors as well as the patient's response at various stages of recovery. The first 48 hrs in hospital, despite being the most resource-intensive period, unfortunately result in the highest mortality. These patients are on life support at the time of their hospital admission and adequate and reliable clinical examination is impossible. Thus, patients receive treatment despite lack of a clear understanding of their prognoses.

Hypothesis: Admission Computed Tomographic Perfusion (CTP) can diagnose brain death reliably in severe TBI patients in early stage upon hospital admission, which is not recognised in the usual clinical practice due to inadequate reliable clinical examination. In a small prospective pilot study of 19 patients with severe TBI, admission CTP could predict early in hospital mortality with 75% sensitivity, 100% specificity, 100% positive predictive value (PPV) and 94% negative predictive value (NPV) and perfect inter-rater reliability (kappa=1). We propose ACT-TBI study to evaluate CTP as a triage tool to diagnose early mortality at the time of admission in patients with severe TBI.

Primary Objective: To validate admission CTP features of brain death, relative to the clinical examination outcome, for characterizing early in-hospital mortality.

Secondary objectives: To establish the safety and interrater reliability of admission CTP.

DETAILED DESCRIPTION:
Objectives of the ACT-TBI study:

In patients with severe TBI,

1. To validate admission CTP features of brain death, relative to the clinical examination outcome, for characterizing early in-hospital mortality.
2. To establish the safety and inter-rater reliability of features of brain death on admission CTP.
3. To evaluate the determinants (age, sex, and GCS score) influencing the variability in response of CTP.
4. To establish the usefulness of CTP in facilitating timely organ transplantation, if possible.

Research Design and Method The ACT-TBI study is a prospective, multi-centre, cohort study in patients with severe TBI and will be conducted in 4 different Canadian centres (Winnipeg, Ottawa, Montreal, and Halifax) over the next 4 years.

Those patients meeting eligibility criteria will be identified by a dedicated research nurse with the help of the trauma team at the time of hospital admission, with the ACT-TBI study protocol will be activated at the time of their first diagnostic imaging. A deferral of consent will be obtained like that in the pilot study.

Clinical Examination- The results of initial clinical, laboratory and imaging assessment will be recorded as per the IMPACT (International Mission for Prognosis and Analysis of Clinical Trials in TBI) core and extended models. The clinical examination will occur during a sedation hold, when possible acknowledging some confounding from effect of residual sedation.

Radiological Examinations Upon hospital admission, at the time of initial diagnostic imaging, besides the standard diagnostic tests of whole-body CT scan, enrolled patients will undergo the whole head imaging protocol with CTP.

Plain computed tomography (CT) of head: As a standard imaging protocol, plain CT of head will be performed for severe TBI patients. These images will be assessed for the presence of various lesions (subarachnoid hemorrhage, sub-dural hemorrhage, epidural hemorrhage, intra-ventricular hemorrhage, cerebral contusions, and edema).

Computed tomography perfusion (CTP): Besides, a standard imaging protocol, CTP imaging protocol for whole head will be performed. Images will be acquired following our previously published protocol. In brief, a total of 40 mL of CT contrast media will be injected at a rate of 5 mL/sec. A set of axial images with a slice thickness of 5 mm for the perfusion analysis will be reconstructed. CTP images will only be acquired. The anonymized images will be transferred and stored in the secured imaging core lab, department of Radiology, University of Manitoba, for processing and interpretation later. CTP will be processed using a semiautomatic deconvolution algorithm on a vendor neutral software package (Oleasphere). CTP will be assessed both quantitatively as well as qualitatively.

* Quantitative assessment: brain death will be defined as Cerebral Blood Flow (CBF) <5 mL/100g/min and Cerebral Blood Volume (CBV) <2 mL/100g in the brainstem.
* Qualitative assessment: brain death will be defined as matched decrease of CBF and CBV in the brainstem. The perfusion maps for CBF and CBV will be assessed for binary outcome of 'dead' or 'not-dead', according to our previously published methods.

The perfusion images will be assessed by the two independent neuroradiologists, who are blinded to the clinical status of the patient and also to each other's assessment. In case of disagreement, the expert neuroradiologist opinion will be employed to have a consensus agreement for the final analysis.

Post-perfusion care: Since the prognostic value of CTP has not been established in patients with severe TBI, the outcomes of CTP will not be made available to the clinical team involved in patient care. All patients will receive the standard care.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Severe head injury with the activation of the trauma code
* GCS score ≤ 8 after initial resuscitation
* On mechanical respiratory ventilation at the time of imaging

Exclusion Criteria:

* No known GCS after initial resuscitation
* Known pregnancy
* Known contraindication to CT contrast agent, e.g.,allergy or anaphylactic reaction
* Known end-stage renal disease stage 4-5 (eGFR < 30 mL/min/1.73 m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome is a binary outcome of mortality ('dead') or survival ('not-dead') in the first 48 hours of hospital admission. | 48 hours
  The primary outcome of this study is determining the mortality ('dead') or survival ('not-dead') in the first 48 hours of hospital admission using CTP.

SECONDARY OUTCOMES:
In-hospital mortality at the end of hospital discharge. | 6 months
  the secondary outcome of this study is to determine In-hospital mortality at the end of hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Jai Shankar, MD FRCPC, Principal Investigator — University of Manitoba; Frederick Zeiler, MD FRCPC, Principal Investigator — University of Manitoba
Locations (4):
- Canada (4):
  - Health Sciences Centre, Winnipeg, Manitoba
  - QEII Health Scienecs Centre, Halifax, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alcock S, Batoo D, Ande SR, Grierson R, Essig M, Martin D, Trivedi A, Sinha N, Leeies M, Zeiler FA, Shankar JJS. Early diagnosis of mortality using admission CT perfusion in severe traumatic brain injury patients (ACT-TBI): protocol for a prospective cohort study. BMJ Open. 2021 Jun 9;11(6):e047305. doi: 10.1136/bmjopen-2020-047305. PMID 34108167